CLINICAL TRIAL: NCT05054010
Title: Identification and Characterization of Commercial RUO Antibodies for the Detection of Specific Breast Cancer Tumoral Markers Expressed in Potential Circulating Tumoral Cells (CTCs)
Brief Title: Identification of Breast Cancer Specific Markers in Patients Compared to Healthy Participants
Status: Active, not recruiting | Type: Observational
Sponsor: Tethis S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: TET-21-001
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer Biomarker; Circulating Tumoral Cell; Immunofluorescence Assay; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early Breast Cancer patients: Early stage breast cancer category is based on the definition of the European Society of medical Oncology and is defined as disease confined to the breast with or without regional lymph node involvement
- Metastatic Breast Cancer patients: Metastatic breast cancer category is based on the definition of the European Society of Medical Oncology and is defined as disease spread to other parts of the body, such as bones, liver or lungs (also called stage IV). Tumours at distant sites are called metastases.
- Healthy donors: Participants who are in good health and without history of cancer disease

SUMMARY:
This is an exploratory research study with the aim of identifying specific cancer biomarkers in various subtypes of breast cancer. Blood samples will be collected from 60 participants divided into 40 patients and 20 healthy donors. An amendment to the research has been proposed to enroll 24 additional participants divided into 12 patients and 12 healthy donors.

DETAILED DESCRIPTION:
In this research study different commercial RUO (Research Use Only) antibodies will be purchased and then tested on blood samples obtained by participants affected by breast cancer and by healthy participants as control. Sixty participants will be enrolled belonging to different categories: 20 participants affected by early breast cancer, 20 participants affected by metastatic breast cancer, and 20 healthy volunteers to be used as negative control.

After signing the informed consent form, participants will be screened to evaluate if they meet the eligibility criteria. If all the criteria are met, participants will be enrolled into the study and will be asked to provide some demographic and other data. A 13 ml blood sample will be collected by the subjects and shipped to Tethis laboratories in order to be processed and analysed.

An amendment has been proposed to enroll 24 additional participants divided into 12 patients and 12 healthy donors. During the amendment, participants will be enrolled to test the analytical capacity of the antibodies evaluated in the first part on samples processed with different methods in order to select the optimal one for future development.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give and sign a written informed consent for participation in the study.
* Female aged 18 years or above.
* Diagnosed with early breast cancer (stage I and II) or metastatic breast cancer.
* Healthy participants who visit the site for reason other than cancer diagnosis (including breast cancer).

Exclusion Criteria:

* History of other malignancies other than breast cancer (for healthy participants includes also breast cancer).
* Undergone surgery or treatment for breast cancer before enrollment (only for early breast cancer).
* Presence of known severe coagulation or haematological disorder
* Known Pregnancy
* Absence of written signed informed consent for participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from among the people who visit the Breast Surgery department
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of commercial Antibodies capable of Identify specific Breast Cancer Biomarkers | 1 day (at the blood draw)
  Qualitative Assessment of Staining Positivity for different Breast Cancer Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Oreste Gentilini, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
This is a basic research study without an IPD information sharing plan

REFERENCES:
- [Background] Hench IB, Hench J, Tolnay M. Liquid Biopsy in Clinical Management of Breast, Lung, and Colorectal Cancer. Front Med (Lausanne). 2018 Jan 30;5:9. doi: 10.3389/fmed.2018.00009. eCollection 2018. PMID 29441349
- [Background] Rawal S, Yang YP, Cote R, Agarwal A. Identification and Quantitation of Circulating Tumor Cells. Annu Rev Anal Chem (Palo Alto Calif). 2017 Jun 12;10(1):321-343. doi: 10.1146/annurev-anchem-061516-045405. Epub 2017 Mar 6. PMID 28301753
- [Background] Carbone R, Marangi I, Zanardi A, Giorgetti L, Chierici E, Berlanda G, Podesta A, Fiorentini F, Bongiorno G, Piseri P, Pelicci PG, Milani P. Biocompatibility of cluster-assembled nanostructured TiO2 with primary and cancer cells. Biomaterials. 2006 Jun;27(17):3221-9. doi: 10.1016/j.biomaterials.2006.01.056. Epub 2006 Feb 28. PMID 16504283
- [Background] Zanardi A, Bandiera D, Bertolini F, Corsini CA, Gregato G, Milani P, Barborini E, Carbone R. Miniaturized FISH for screening of onco-hematological malignancies. Biotechniques. 2010 Jul;49(1):497-504. doi: 10.2144/000113445. PMID 20615202
- [Background] Krol I, Schwab FD, Carbone R, Ritter M, Picocci S, De Marni ML, Stepien G, Franchi GM, Zanardi A, Rissoglio MD, Covelli A, Guidi G, Scarinci D, Castro-Giner F, Mazzarella L, Doglioni C, Borghi F, Milani P, Kurzeder C, Weber WP, Aceto N. Detection of clustered circulating tumour cells in early breast cancer. Br J Cancer. 2021 Jul;125(1):23-27. doi: 10.1038/s41416-021-01327-8. Epub 2021 Mar 24. PMID 33762721
- [Background] Aceto N, Bardia A, Wittner BS, Donaldson MC, O'Keefe R, Engstrom A, Bersani F, Zheng Y, Comaills V, Niederhoffer K, Zhu H, Mackenzie O, Shioda T, Sgroi D, Kapur R, Ting DT, Moy B, Ramaswamy S, Toner M, Haber DA, Maheswaran S. AR Expression in Breast Cancer CTCs Associates with Bone Metastases. Mol Cancer Res. 2018 Apr;16(4):720-727. doi: 10.1158/1541-7786.MCR-17-0480. Epub 2018 Feb 16. PMID 29453314
- [Background] Xu L, Jia S, Li H, Yu Y, Liu G, Wu Y, Liu X, Liu C, Zhou Y, Zhang Z, Sheng Y. Characterization of circulating tumor cells in newly diagnosed breast cancer. Oncol Lett. 2018 Feb;15(2):2522-2528. doi: 10.3892/ol.2017.7540. Epub 2017 Dec 6. PMID 29434968
- [Background] Fujii T, Reuben JM, Huo L, Espinosa Fernandez JR, Gong Y, Krupa R, Suraneni MV, Graf RP, Lee J, Greene S, Rodriguez A, Dugan L, Louw J, Lim B, Barcenas CH, Marx AN, Tripathy D, Wang Y, Landers M, Dittamore R, Ueno NT. Androgen receptor expression on circulating tumor cells in metastatic breast cancer. PLoS One. 2017 Sep 28;12(9):e0185231. doi: 10.1371/journal.pone.0185231. eCollection 2017. PMID 28957377